CLINICAL TRIAL: NCT05791565
Title: A Single Dose Two-way Cross-over Study in Healthy Participants to Compare the Pharmacokinetics (PK) of Salbutamol Administered Via Metered Dose Inhalers Containing Propellants HFA-152a and HFA-134a
Brief Title: Green (Sustainable) VENTOLIN - Pharmacokinetics (PK) Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 219430
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Asthma
Keywords: Cross-over; Healthy volunteers; Salbutamol; Pharmacokinetics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This is a 2-way cross-over study.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salbutamol HFA-152a MDI followed by Salbutamol HFA-134a MDI (Experimental): Participants will receive Salbutamol HFA-152a MDI in treatment period 1 followed by Salbutamol HFA-134a MDI in treatment period 2. There will be a minimum washout period of 72 hours between each treatment period.
  Interventions: Drug: Salbutamol HFA-152a; Drug: Salbutamol HFA-134a
- Salbutamol HFA-134a MDI followed by Salbutamol HFA-152a MDI (Experimental): Participants will receive Salbutamol HFA-134a MDI in treatment period 1 followed by Salbutamol HFA-152a MDI in treatment period 2. There will be a minimum washout period of 72 hours between each treatment period.
  Interventions: Drug: Salbutamol HFA-152a; Drug: Salbutamol HFA-134a

INTERVENTIONS:
Drug: Salbutamol HFA-152a — Salbutamol HFA-152a will be administered.
Drug: Salbutamol HFA-134a — Salbutamol HFA-134a will be administered.

SUMMARY:
This study will be conducted to compare the PK of salbutamol administered via metered dose inhalers (MDI) containing propellants 1,1-difluroethane (HFA-152a) and 1,1,1,2-tetrafluoroethane (HFA-134a) in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 55 years, inclusive, at screening
* Body mass index 18.0 to 30.0 kilograms per meter square (kg/m^2), inclusive, at screening
* Weight: greater than or equal to (>=)50 kg
* At screening, females must not be pregnant or lactating, or of non-childbearing potential
* Female participants of childbearing potential who have a fertile male sexual partner must agree to use adequate contraception
* Male participants, if not surgically sterilized, must agree to use adequate contraception
* Good physical and mental health on the basis of medical history, physical examination, clinical laboratory, electrocardiogram, and vital signs, as judged by the investigator
* Willing and able to sign the informed consent form

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data
* History or presence of any form of asthma, including childhood asthma and exercise induced asthma
* Current enrollment or past participation in this clinical study
* Participants with clinically significant abnormalities
* A positive pre-study drug/alcohol screen or a history (or suspected history) of alcohol misuse or substance abuse
* Positive nasopharyngeal polymerase chain reaction test for severe acute respiratory syndrome-corona virus type 2 (SARS-CoV-2) on Day -1 or any known close contact with a person who tested positive for SARS-CoV-2 or with a coronavirus disease 2019 participant within 2 weeks prior to admission
* Impairment which would prevent the correct and consistent use of an MDI, as determined by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Groups:
- Salbutamol HFA-152a MDI Followed by Salbutamol HFA-134a MDI: Healthy participants received Salbutamol Hydrofluoroalkane (HFA)-152a metered dose inhaler (MDI) suspension as a single 800 µg (8 x 100 µg dose at 20-second intervals) inhalation on Day 1 of treatment period 1. In treatment period 2, participants received Salbutamol HFA-134a MDI suspension as a single 800 µg (8 x 100 µg dose at 20-second intervals) inhalation on Day 4. There was a minimum washout period of 72 hours between each treatment period.
- Salbutamol HFA-134a MDI Followed by Salbutamol HFA-152a MDI: Healthy participants received Salbutamol Hydrofluoroalkane (HFA)-134a metered dose inhaler (MDI) suspension as a single 800 µg (8 x 100 µg dose at 20-second intervals) inhalation on Day 1 of treatment period 1. In treatment period 2, Salbutamol HFA-152a MDI suspension as a single 800 µg (8 x 100 µg dose at 20-second intervals) via inhalation on Day 4. There was a minimum washout period of 72 hours between each treatment period.
Period: Period 1 (Day 1)
Arm/Group | Salbutamol HFA-152a MDI Followed by Salbutamol HFA-134a MDI | Salbutamol HFA-134a MDI Followed by Salbutamol HFA-152a MDI
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout Period (Minimum 72 Hours)
Arm/Group | Salbutamol HFA-152a MDI Followed by Salbutamol HFA-134a MDI | Salbutamol HFA-134a MDI Followed by Salbutamol HFA-152a MDI
Started | 14 | 14
Completed | 13 | 14
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2 (Day 4)
Arm/Group | Salbutamol HFA-152a MDI Followed by Salbutamol HFA-134a MDI | Salbutamol HFA-134a MDI Followed by Salbutamol HFA-152a MDI
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Salbutamol HFA-152a MDI Followed by Salbutamol HFA-134a MDI | Salbutamol HFA-134a MDI Followed by Salbutamol HFA-152a MDI | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.4 (11.03) | 31.5 (11.59) | 31.5 (11.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 5 | 9 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve up to 30 Minutes Post-dose (AUC (0-30 Min)) of Salbutamol
Description: Blood samples were collected for pharmacokinetic (PK) analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose and post dose 3, 5, 10, 15, 20 and 30 minutes on Day 1 and Day 4
Population: Pharmacokinetic population included all participants in the safety population who received at least one dose of study treatment and had at least one non-missing PK assessment. Only those participants with data available at specified time points have been analyzed. 1 participant in Salbutamol HFA-152a MDI arm had out of window samples resulting in two samples with the same collection time. Therefore, data could not be calculated and were excluded from the analysis.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hour*nanogram/milliliter (h*ng/mL)
Groups:
- Salbutamol HFA-152a MDI: Healthy participants received a single dose of 800 µg (8 x 100 µg dose at 20-second intervals) Salbutamol HFA-152a MDI suspension as inhalation on Day 1 or Day 4 (in either treatment Period 1 or 2).
- Salbutamol HFA-134a MDI: Healthy participants received a single dose of 800 µg (8 x 100 µg dose at 20-second intervals) Salbutamol HFA-134a MDI suspension as inhalation on Day 1 or Day 4 (in either treatment Period 1 or 2).
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 27 | 27
Hour*nanogram/milliliter (h*ng/mL) | 0.622 [0.535 to 0.724] | 0.536 [0.461 to 0.623]
Statistical Analysis 1: Comparison: Salbutamol HFA-152a MDI vs Salbutamol HFA-134a MDI; Test type: Other; Ratio of Geometric LS Means = 1.1609, 90% CI 2-sided [1.0221 to 1.3185] — Ratio of the Geometric LS means = Geometric LS mean of the Salbutamol HFA-152a MDI to the Geometric LS mean of the Salbutamol HFA-134a MDI

2. Primary Outcome: AUC From Time 0 to Infinity (AUC[0-inf]) of Salbutamol
Description: as for outcome 1
Time Frame: Pre-dose and post dose 0.05, 0.08, 0.17, 0.25, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 hours on Day 1 and Day 4
Population: as for outcome 1
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 27 | 27
Hour*nanogram/milliliter (h*ng/mL) | 21.1 [19.7 to 22.6] | 15.0 [14.0 to 16.1]
Statistical Analysis 1: Comparison: Salbutamol HFA-152a MDI vs Salbutamol HFA-134a MDI; Test type: Other; Ratio of the Geometric LS Means = 1.4081, 90% CI 2-sided [1.2998 to 1.5255] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC From Time 0 to Time t (AUC[0-t]) of Salbutamol
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hour*nanogram/millilitre (h*ng/mL)
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 27 | 27
Hour*nanogram/millilitre (h*ng/mL) | 19.0 [17.7 to 20.5] | 13.7 [12.7 to 14.7]
Statistical Analysis 1: Comparison: Salbutamol HFA-152a MDI vs Salbutamol HFA-134a MDI; Test type: Other; Ratio of the Geometric LS Means = 1.3885, 90% CI 2-sided [1.2793 to 1.5070] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Salbutamol
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: nanogram/millilitre (ng/mL)
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 27 | 27
nanogram/millilitre (ng/mL) | 2.36 [2.15 to 2.60] | 1.80 [1.63 to 1.97]
Statistical Analysis 1: Comparison: Salbutamol HFA-152a MDI vs Salbutamol HFA-134a MDI; Test type: Other; Ratio of the Geometric LS Means = 1.3141, 90% CI 2-sided [1.1816 to 1.4614] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Time to Cmax (Tmax) of Salbutamol
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 27 | 27
hour (h) | 2.00 [0.33 to 5.00] | 1.50 [0.05 to 4.00]

6. Secondary Outcome: Apparent Terminal Phase Half-life (t1/2) of Salbutamol
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 27 | 27
hour (h) | 7.650 (21.1) | 7.297 (17.1)

7. Secondary Outcome: Minimum Observed Serum Potassium Level (Emin, K) After Dosing of Salbutamol
Description: Minimum observed concentration of potassium levels after dose are presented.
Time Frame: 0.25, 0.5, 1, 1.5, 2 and 4 hours post-dose on each dosing day (Days 1 and 4)
Population: Pharmacodynamic population included all participants who received at least one dose of study intervention and have at least one non-missing potassium concentration result. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: millimoles per liter (mmol/L)
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 28 | 27
millimoles per liter (mmol/L) | 3.94 [3.884 to 4.003] | 3.96 [3.902 to 4.023]

8. Secondary Outcome: Weighted Mean Serum Potassium (0-4 Hour) (AUEC, K)
Description: Weighed mean of serum potassium was calculated as summation of each interval. Each interval calculated as: (C2-C1)/2 * (t2-t1), where C2 and t2 are serum potassium and timepoint at the end of each interval, and C1 and t1 are serum potassium and timepoint at the start of each interval.
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2 and 4 hours post-dose on each dosing day (Days 1 and 4)
Population: Pharmacodynamic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: millimoles per liter (mmol/L)
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 28 | 27
millimoles per liter (mmol/L) | 4.15 [4.086 to 4.213] | 4.17 [4.110 to 4.240]

9. Secondary Outcome: Maximum Observed Heart Rate (Emax, HR) After Dosing of Salbutamol
Description: Maximum observed heart rate (HR) after dose is presented.
Time Frame: 0.25, 0.5, 1, 1.5, 2 and 4 hours post-dose on each dosing day (Days 1 and 4)
Population: Pharmacodynamic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Beats per minute (beats/min)
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 28 | 27
Beats per minute (beats/min) | 74.2 [71.25 to 77.35] | 73.4 [70.43 to 76.50]

10. Secondary Outcome: Weighted Mean Heart Rate (0-4 Hour) (AUEC, HR)
Description: Weighed mean of HR was calculated as summation of each interval. Each interval calculated as: (C2-C1)/2 * (t2-t1), where C2 and t2 are HR and timepoint at the end of each interval, and C1 and t1 are HR and timepoint at the start of each interval.
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2 and 4 hours post-dose on each dosing day (Days 1 and 4)
Population: Pharmacodynamic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Beats per minute (beats/min)
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 28 | 27
Beats per minute (beats/min) | 61.4 [58.99 to 63.91] | 60.9 [58.51 to 63.41]

11. Secondary Outcome: Maximum Observed QTcF (Emax, QTcF) After Dosing of Salbutamol
Description: Maximum observed QTcF after dose are presented.
Time Frame: 0.25, 0.5, 1, 1.5, 2 and 4 hours post-dose on each dosing day (Days 1 and 4)
Population: Pharmacodynamic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 28 | 27
Milliseconds | 408.7 [403.34 to 414.14] | 405.5 [400.15 to 410.90]

12. Secondary Outcome: Weighted Mean QTcF (0-4 Hour) (AUEC, QTcF)
Description: Weighed mean of QTcF was calculated as summation of each interval. Each interval calculated as: [(C2+C1)/2×(t2-t1)]/Total time (Tlast-Tfirst, ie 4-0 hour) where C2 and t2 are concentration and timepoint at the end of each interval, and C1 and t1 are concentration and timepoint at the start of each interval. Tlast is the end of the last collection interval, and Tfirst is the start of the first collection interval.
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2 and 4 hours post-dose on each dosing day (Days 1 and 4)
Population: Pharmacodynamic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 28 | 27
Milliseconds | 384.6 [380.01 to 389.29] | 380.8 [376.19 to 385.41]

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A TEAE is an event that emerges during treatment having been absent pre-treatment or worsens relative to the pre-treatment state. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity or is a congenital anomaly/birth defect. A summary of number of participants with any AEs and SAEs are presented. AEs were coded using the Medical Dictionary for Regulatory Affairs (MedDRA dictionary).
Time Frame: Up to 5 days
Population: Safety population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 28 | 27
Participants
  Any TEAEs | 9 | 7
  Any SAEs | 0 | 0

14. Secondary Outcome: Absolute Values of Electrocardiogram (ECG) Parameters: PR Interval, QRS Duration, QT Interval and Corrected QT (QTc) Interval
Description: A standard 12-lead ECG was obtained using an ECG machine that automatically calculates the HR and measures PR, QRS, QT, and QTcF intervals. The ECG was obtained after the participant has been resting for at least 5 minutes in the supine position. Pre-dose 12-lead ECG was measured in triplicate. The 3 pre-dose measures was averaged for QTc interval and HR to derive one baseline value. Each individual capture of the triplicate 12-lead ECG set was separated by 1 to 5 minutes between the first and the third ECG. Baseline is defined as the last observation recorded before the first study drug administration in each dosing period.
Time Frame: Baseline (Pre-dose at Day 1 and Day 4); 0.25, 0.5, 1 hour (h), 1.5 h, 2 h, 4 h post-dose at Day 1 and Day 4
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Milliseconds
  PR, Baseline (Day 1, Predose) | 160.5 (25.47) | 157.1 (17.57)
  PR, Day 1, 15 min post-dose | 149.2 (21.93) | 150.2 (16.59)
  PR, Day 1, 30 min post-dose | 149.8 (23.13) | 153.2 (17.12)
  PR, Day 1, 1 h post-dose | 151.6 (20.25) | 151.4 (17.05)
  PR, Day 1, 1.5 h post-dose | 153.2 (22.04) | 154.6 (16.99)
  PR, Day 1, 2 h post-dose | 156.2 (23.40) | 153.5 (18.47)
  PR, Day 1, 4 h post-dose | 153.3 (24.82) | 154.4 (16.40)
  PR, Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  PR, Baseline (Day 4, Predose) | 157.6 (18.16) | 159.1 (24.95)
  PR, Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  PR, Day 4, 15 min post-dose | 147.5 (17.17) | 146.6 (22.61)
  PR, Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  PR, Day 4, 30 min post-dose | 151.4 (17.08) | 151.1 (25.81)
  PR, Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  PR, Day 4, 1 h post-dose | 150.2 (15.34) | 153.8 (24.73)
  PR, Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  PR, Day 4, 1.5 h post-dose | 153.6 (17.91) | 154.9 (21.45)
  PR, Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  PR, Day 4, 2 h post-dose | 149.3 (18.03) | 153.4 (22.01)
  PR, Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  PR, Day 4, 4 h post-dose | 152.3 (18.51) | 157.7 (25.82)
  QRS duration, Baseline (Day 1, Predose) | 93.0 (9.27) | 98.5 (9.18)
  QRS duration, Day 1, 15 min post-dose | 92.0 (8.73) | 98.8 (10.28)
  QRS duration, Day 1, 30 min post-dose | 92.1 (9.68) | 97.6 (11.97)
  QRS duration, Day 1, 1 h post-dose | 91.5 (9.98) | 97.6 (10.44)
  QRS duration, Day 1, 1.5 h post-dose | 92.4 (8.87) | 97.0 (10.91)
  QRS duration, Day 1, 2 h post-dose | 92.1 (8.12) | 99.4 (9.87)
  QRS duration, Day 1, 4 h post-dose | 91.8 (7.95) | 98.0 (8.82)
  QRS duration, Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  QRS duration, Baseline (Day 4, Predose) | 97.9 (8.99) | 92.4 (7.78)
  QRS duration, Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, Day 4, 15 min post-dose | 96.9 (9.56) | 91.4 (7.41)
  QRS duration, Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, Day 4, 30 min post-dose | 97.6 (9.58) | 91.6 (8.28)
  QRS duration, Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, Day 4, 1 h post-dose | 96.6 (9.04) | 92.2 (8.51)
  QRS duration, Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, Day 4, 1.5 h post-dose | 96.2 (11.45) | 92.6 (7.02)
  QRS duration, Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, Day 4, 2 h post-dose | 97.3 (8.92) | 93.2 (7.96)
  QRS duration, Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, Day 4, 4 h post-dose | 96.3 (9.12) | 90.2 (8.12)
  QT interval, Baseline (Day 1, Predose) | 404.2 (27.19) | 398.3 (19.86)
  QT interval, Day 1, 15 min post-dose | 374.9 (26.22) | 372.5 (18.15)
  QT interval, Day 1, 30 min post-dose | 377.2 (27.45) | 380.8 (21.76)
  QT interval, Day 1, 1 h post-dose | 386.7 (26.95) | 384.1 (23.81)
  QT interval, Day 1, 1.5 h post-dose | 393.9 (24.80) | 385.3 (22.84)
  QT interval, Day 1, 2 h post-dose | 399.4 (25.22) | 391.2 (23.68)
  QT interval, Day 1, 4 h post-dose | 407.8 (27.67) | 395.7 (23.27)
  QT interval, Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  QT interval, Baseline (Day 4, Predose) | 400.8 (22.66) | 403.5 (25.28)
  QT interval, Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  QT interval, Day 4, 15 min post-dose | 373.8 (18.52) | 374.2 (22.98)
  QT interval, Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  QT interval, Day 4, 30 min post-dose | 379.0 (19.41) | 379.8 (22.75)
  QT interval, Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  QT interval, Day 4, 1 h post-dose | 382.8 (20.18) | 386.2 (19.16)
  QT interval, Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  QT interval, Day 4, 1.5 h post-dose | 386.7 (20.72) | 388.5 (20.27)
  QT interval, Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  QT interval, Day 4, 2 h post-dose | 393.0 (20.55) | 395.5 (18.59)
  QT interval, Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  QT interval, Day 4, 4 h post-dose | 397.0 (22.25) | 405.4 (22.90)
  QTc interval, Baseline (Day 1, Predose) | 402.1 (15.47) | 404.2 (14.33)
  QTc interval, Day 1, 15 min post-dose | 396.9 (21.86) | 397.1 (12.97)
  QTc interval, Day 1, 30 min post-dose | 399.6 (19.47) | 400.1 (14.56)
  QTc interval, Day 1, 1 h post-dose | 400.6 (20.43) | 398.9 (14.45)
  QTc interval, Day 1, 1.5 h post-dose | 401.9 (18.11) | 399.9 (12.09)
  QTc interval, Day 1, 2 h post-dose | 402.4 (16.10) | 396.8 (13.55)
  QTc interval, Day 1, 4 h post-dose | 403.2 (19.19) | 403.1 (13.57)
  QTc interval, Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  QTc interval, Baseline (Day 4, Predose) | 402.2 (14.44) | 397.4 (16.30)
  QTc interval, Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, Day 4, 15 min post-dose | 398.0 (15.00) | 396.3 (18.45)
  QTc interval, Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, Day 4, 30 min post-dose | 402.0 (14.22) | 398.2 (23.29)
  QTc interval, Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, Day 4, 1 h post-dose | 399.2 (17.52) | 398.8 (17.62)
  QTc interval, Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, Day 4, 1.5 h post-dose | 397.9 (15.28) | 392.7 (19.45)
  QTc interval, Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, Day 4, 2 h post-dose | 402.9 (16.16) | 397.8 (17.85)
  QTc interval, Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, Day 4, 4 h post-dose | 402.1 (18.19) | 398.2 (16.22)

15. Secondary Outcome: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval and QTc Interval
Description: A standard 12-lead ECG was obtained using an ECG machine that automatically calculates the HR and measures PR, QRS, QT, and QTcF intervals. The ECG was obtained after the participant has been resting for at least 5 minutes in the supine position. Pre-dose 12-lead ECG was measured in triplicate. The 3 pre-dose measures was averaged for QTc interval and HR to derive one baseline value. Each individual capture of the triplicate 12-lead ECG set was separated by 1 to 5 minutes between the first and the third ECG. Screening and post-dose 12-lead ECG measurements were single measurements.
Time Frame: Baseline (Pre-dose at Day 1 and Day 4); 0.25, 0.5, 1 hour (h), 1.5 h, 2 h, 4 h post-dose at Day 1 and Day 4
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Milliseconds
  PR, Baseline (Day 1, Predose) | 160.5 (25.47) | 157.1 (17.57)
  PR, CFB to Day 1, 15 min post-dose | -11.3 (11.74) | -6.9 (7.00)
  PR, CFB to Day 1, 30 min post-dose | -10.7 (11.67) | -3.9 (5.14)
  PR, CFB to Day 1, 1 h post-dose | -8.9 (13.32) | -5.6 (7.23)
  PR, CFB to Day 1, 1.5 h post-dose | -7.3 (9.61) | -2.5 (6.72)
  PR, CFB to Day 1, 2 h post-dose | -4.3 (5.62) | -3.6 (8.06)
  PR, CFB to Day 1, 4 h post-dose | -7.2 (6.57) | -2.6 (5.06)
  PR, Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  PR, Baseline (Day 4, Predose) | 157.6 (18.16) | 159.1 (24.95)
  PR, CFB to Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  PR, CFB to Day 4, 15 min post-dose | -10.1 (12.11) | -12.5 (9.37)
  PR, CFB to Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  PR, CFB to Day 4, 30 min post-dose | -6.2 (8.05) | -8.0 (8.10)
  PR, CFB to Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  PR, CFB to Day 4, 1 h post-dose | -7.4 (11.19) | -5.3 (6.46)
  PR, CFB to Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  PR, CFB to Day 4, 1.5 h post-dose | -4.0 (9.46) | -4.2 (7.73)
  PR, CFB to Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  PR, CFB to Day 4, 2 h post-dose | -8.4 (12.49) | -5.7 (5.59)
  PR, CFB to Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  PR, CFB to Day 4, 4 h post-dose | -5.4 (10.65) | -1.4 (2.50)
  QRS duration, Baseline (Day 1, Predose) | 93.0 (9.27) | 98.5 (9.18)
  QRS duration, CFB to Day 1, 15 min post-dose | -1.0 (3.72) | 0.3 (4.07)
  QRS duration, CFB to Day 1, 30 min post-dose | -0.9 (4.04) | -0.9 (5.37)
  QRS duration, CFB to Day 1, 1 h post-dose | -1.5 (3.25) | -0.9 (4.37)
  QRS duration, CFB to Day 1, 1.5 h post-dose | -0.6 (3.59) | -1.5 (4.72)
  QRS duration, CFB to Day 1, 2 h post-dose | -0.9 (5.90) | 0.9 (5.05)
  QRS duration, CFB to Day 1, 4 h post-dose | -1.2 (4.49) | -0.5 (3.88)
  QRS duration, Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  QRS duration, Baseline (Day 4, Predose) | 97.9 (8.99) | 92.4 (7.78)
  QRS duration, CFB to Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, CFB to Day 4, 15 min post-dose | -1.0 (5.43) | -1.0 (2.92)
  QRS duration, CFB to Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, CFB to Day 4, 30 min post-dose | -0.2 (4.66) | -0.8 (2.42)
  QRS duration, CFB to Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, CFB to Day 4, 1 h post-dose | -1.2 (5.54) | -0.2 (3.03)
  QRS duration, CFB to Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, CFB to Day 4, 1.5 h post-dose | -1.6 (5.72) | 0.2 (3.27)
  QRS duration, CFB to Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, CFB to Day 4, 2 h post-dose | -0.6 (5.76) | 0.8 (2.52)
  QRS duration, CFB to Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  QRS duration, CFB to Day 4, 4 h post-dose | -1.6 (4.45) | -2.2 (4.68)
  QT interval, Baseline (Day 1, Predose) | 404.2 (27.19) | 398.3 (19.86)
  QT interval, CFB to Day 1, 15 min post-dose | -29.4 (21.45) | -25.8 (9.94)
  QT interval, CFB to Day 1, 30 min post-dose | -27.0 (20.03) | -17.5 (12.43)
  QT interval, CFB to Day 1, 1 h post-dose | -17.5 (11.76) | -14.2 (13.22)
  QT interval, CFB to Day 1, 1.5 h post-dose | -10.3 (13.93) | -13.0 (12.35)
  QT interval, CFB to Day 1, 2 h post-dose | -4.9 (17.13) | -7.1 (12.43)
  QT interval, CFB to Day 1, 4 h post-dose | 3.6 (14.90) | -2.6 (15.25)
  QT interval, Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  QT interval, Baseline (Day 4, Predose) | 400.8 (22.66) | 403.5 (25.28)
  QT interval, CFB to Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  QT interval, CFB to Day 4, 15 min post-dose | -27.0 (11.08) | -29.2 (11.67)
  QT interval, CFB to Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  QT interval, CFB to Day 4, 30 min post-dose | -21.8 (10.66) | -23.6 (7.61)
  QT interval, CFB to Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  QT interval, CFB to Day 4, 1 h post-dose | -18.0 (10.77) | -17.3 (12.08)
  QT interval, CFB to Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  QT interval, CFB to Day 4, 1.5 h post-dose | -14.1 (9.27) | -15.0 (10.79)
  QT interval, CFB to Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  QT interval, CFB to Day 4, 2 h post-dose | -7.8 (9.43) | -8.0 (12.90)
  QT interval, CFB to Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  QT interval, CFB to Day 4, 4 h post-dose | -3.8 (12.70) | 1.9 (11.72)
  QTc interval, Baseline (Day 1, Predose) | 402.1 (15.47) | 404.2 (14.33)
  QTc interval, CFB to Day 1, 15 min post-dose | -5.1 (21.16) | -7.1 (6.37)
  QTc interval, CFB to Day 1, 30 min post-dose | -2.5 (17.30) | -4.1 (6.80)
  QTc interval, CFB to Day 1, 1 h post-dose | -1.4 (10.95) | -5.4 (7.11)
  QTc interval, CFB to Day 1, 1.5 h post-dose | -0.2 (7.17) | -4.4 (8.30)
  QTc interval, CFB to Day 1, 2 h post-dose | 0.3 (9.79) | -7.4 (7.76)
  QTc interval, CFB to Day 1, 4 h post-dose | 1.1 (8.63) | -1.1 (7.68)
  QTc interval, Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  QTc interval, Baseline (Day 4, Predose) | 402.2 (14.44) | 397.4 (16.30)
  QTc interval, CFB to Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, CFB to Day 4, 15 min post-dose | -4.2 (10.18) | -1.1 (9.09)
  QTc interval, CFB to Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, CFB to Day 4, 30 min post-dose | -0.2 (7.51) | 0.8 (9.81)
  QTc interval, CFB to Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, CFB to Day 4, 1 h post-dose | -3.0 (10.69) | 1.5 (6.15)
  QTc interval, CFB to Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, CFB to Day 4, 1.5 h post-dose | -4.3 (8.74) | -4.7 (6.24)
  QTc interval, CFB to Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, CFB to Day 4, 2 h post-dose | 0.7 (9.56) | 0.4 (6.21)
  QTc interval, CFB to Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  QTc interval, CFB to Day 4, 4 h post-dose | -0.1 (10.27) | 0.8 (4.27)

16. Secondary Outcome: Absolute Values of ECG Parameter: Heart Rate
Description: as for outcome 15
Time Frame: Baseline (Pre-dose at Day 1 and Day 4); 0.25, 0.5, 1 hour (h), 1.5 h, 2 h, 4 h post-dose at Day 1 and Day 4
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Beats per minute
  Baseline (Day 1, Predose) | 59.9 (10.01) | 63.2 (8.12)
  Day 1, 15 min post-dose | 71.6 (8.73) | 73.3 (9.51)
  Day 1, 30 min post-dose | 71.9 (9.98) | 70.5 (11.80)
  Day 1, 1 h post-dose | 67.4 (8.54) | 67.9 (10.86)
  Day 1, 1.5 h post-dose | 63.9 (6.20) | 67.9 (9.34)
  Day 1, 2 h post-dose | 61.5 (6.55) | 63.1 (8.98)
  Day 1, 4 h post-dose | 58.4 (7.32) | 63.9 (9.38)
  Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  Baseline (Day 4, Predose) | 61.1 (8.65) | 57.8 (9.53)
  Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 15 min post-dose | 72.5 (7.14) | 71.8 (11.16)
  Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 30 min post-dose | 72.1 (10.05) | 69.6 (9.89)
  Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 1 h post-dose | 68.6 (9.74) | 66.2 (7.80)
  Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 1.5 h post-dose | 65.9 (9.54) | 62.4 (8.43)
  Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 2 h post-dose | 65.0 (7.84) | 61.2 (7.84)
  Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 4 h post-dose | 62.7 (8.53) | 57.1 (7.95)

17. Secondary Outcome: Change From Baseline in ECG Parameters: Heart Rate
Description: as for outcome 15
Time Frame: Baseline (Pre-dose at Day 1 and Day 4); 0.25, 0.5, 1 hour (h), 1.5 h, 2 h, 4 h post-dose at Day 1 and Day 4
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Beats per minute
  Baseline (Day 1, Predose) | 59.9 (10.01) | 63.2 (8.12)
  CFB Day 1, 15 min post-dose | 11.7 (5.61) | 10.1 (6.45)
  CFB Day 1, 30 min post-dose | 12.0 (5.35) | 7.3 (8.06)
  CFB Day 1, 1 h post-dose | 7.4 (5.37) | 4.7 (7.66)
  CFB Day 1, 1.5 h post-dose | 3.9 (6.64) | 4.7 (6.67)
  CFB Day 1, 2 h post-dose | 1.6 (7.87) | -0.1 (6.28)
  CFB Day 1, 4 h post-dose | -1.6 (6.05) | 0.6 (7.66)
  Baseline (Day 4, Predose) | 61.1 (8.65) | 57.8 (9.53)
  CFB Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  CFB Day 4, 15 min post-dose | 11.4 (4.64) | 14.1 (7.03)
  CFB Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  CFB Day 4, 30 min post-dose | 11.0 (6.63) | 11.8 (5.46)
  CFB Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  CFB Day 4, 1 h post-dose | 7.5 (5.63) | 8.5 (5.58)
  CFB Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  CFB Day 4, 1.5 h post-dose | 4.9 (4.82) | 4.6 (4.46)
  CFB Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  CFB Day 4, 2 h post-dose | 3.9 (4.36) | 3.5 (5.80)
  CFB Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  CFB Day 4, 4 h post-dose | 1.6 (5.89) | -0.7 (5.36)

18. Secondary Outcome: Absolute Values of Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelet Count
Description: Blood samples were collected for analyzing absolute values of Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelet count.
Time Frame: On Day -1 (admission) and Day 5 (Discharge)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Giga cells per liter
  Basophils, Day -1 | 0.03 (0.047) | 0.02 (0.037)
  Basophils, Day 5: number analyzed (Participants) | 14 | 13
  Basophils, Day 5 | 0.01 (0.029) | 0.00 (0.000)
  Eosinophils, Day -1 | 0.16 (0.160) | 0.15 (0.142)
  Eosinophils, Day 5: number analyzed (Participants) | 14 | 13
  Eosinophils, Day 5 | 0.15 (0.094) | 0.18 (0.124)
  Lymphocytes, Day -1 | 2.02 (0.699) | 2.08 (0.471)
  Lymphocytes, Day 5: number analyzed (Participants) | 14 | 13
  Lymphocytes, Day 5 | 1.90 (0.367) | 1.83 (0.477)
  Monocytes, Day -1 | 0.43 (0.133) | 0.42 (0.107)
  Monocytes, Day 5: number analyzed (Participants) | 14 | 13
  Monocytes, Day 5 | 0.36 (0.116) | 0.37 (0.118)
  Neutrophils, Day -1 | 4.46 (1.540) | 4.24 (1.117)
  Neutrophils, Day 5: number analyzed (Participants) | 14 | 13
  Neutrophils, Day 5 | 3.20 (0.954) | 3.15 (0.996)
  Platelet count, Day -1 | 257.07 (62.390) | 247.64 (45.865)
  Platelet count, Day 5: number analyzed (Participants) | 14 | 13
  Platelet count, Day 5 | 235.50 (37.293) | 239.85 (55.306)

19. Secondary Outcome: Absolute Values of Hematology Parameter: Red Blood Cell (RBC) and Reticulocytes Count
Description: Blood samples were collected for analyzing absolute values of red blood cell (RBC) and reticulocytes count.
Time Frame: On Day -1 (admission) and Day 5 (Discharge)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Trillion cells per liter
  RBC, Day -1 | 4.889 (0.3357) | 5.074 (0.5315)
  RBC, Day 5: number analyzed (Participants) | 14 | 13
  RBC, Day 5 | 4.703 (0.5065) | 4.590 (0.2988)
  Reticulocytes, Day -1 | 0.064 (0.0145) | 0.074 (0.0179)
  Reticulocytes, Day 5: number analyzed (Participants) | 14 | 13
  Reticulocytes, Day 5 | 0.073 (0.0159) | 0.065 (0.0127)

20. Secondary Outcome: Absolute Values of Hematology Parameter: Mean Corpuscular Volume (MCV)
Description: Blood samples were collected for analyzing absolute values of Mean Corpuscular Volume (MCV).
Time Frame: On Day -1 (admission) and Day 5 (Discharge)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Femtoliters
  Day -1 | 85.07 (4.009) | 86.14 (4.435)
  Day 5: number analyzed (Participants) | 14 | 13
  Day 5 | 86.50 (4.053) | 85.38 (4.273)

21. Secondary Outcome: Absolute Values of Hematology Parameter: Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected for analyzing absolute values of Mean corpuscular hemoglobin (MCH).
Time Frame: On Day -1 (admission) and Day 5 (Discharge)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Picograms
  Day -1 | 29.453 (1.6398) | 29.832 (1.7107)
  Day 5: number analyzed (Participants) | 14 | 13
  Day 5 | 30.063 (1.6244) | 29.288 (1.8080)

22. Secondary Outcome: Absolute Values of Hematology Parameter: Hemoglobin
Description: Blood samples were collected for analyzing absolute values of Hemoglobin.
Time Frame: On Day -1 (admission) and Day 5 (Discharge)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Grams per Liter
  Day -1 | 143.87 (11.978) | 150.79 (11.125)
  Day 5: number analyzed (Participants) | 14 | 13
  Day 5 | 140.76 (11.437) | 134.35 (11.602)

23. Secondary Outcome: Absolute Values of Hematology Parameter: Hematocrit
Description: Blood samples were collected for analyzing absolute values of Hematocrit.
Time Frame: On Day -1 (admission) and Day 5 (Discharge)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Percentage
  Day -1 | 0.416 (0.0352) | 0.436 (0.0313)
  Day 5: number analyzed (Participants) | 14 | 13
  Day 5 | 0.404 (0.0330) | 0.392 (0.0302)

24. Secondary Outcome: Absolute Values of Clinical Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Creatine Phosphokinase (CPK)
Description: Blood samples were collected for analyzing absolute values of Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Aspartate aminotransferase (AST) and Creatine Phosphokinase (CPK).
Time Frame: On Day -1 (admission) and Day 5 (Discharge)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
International units per Liter
  ALT, Day -1 | 24.21 (13.634) | 24.14 (11.481)
  ALT, Day 5: number analyzed (Participants) | 14 | 13
  ALT, Day 5 | 26.36 (12.959) | 24.38 (14.728)
  ALP, Day -1 | 69.57 (20.429) | 66.36 (19.262)
  ALP, Day 5: number analyzed (Participants) | 14 | 13
  ALP, Day 5 | 61.93 (18.898) | 61.46 (20.206)
  AST, Day -1 | 17.64 (10.725) | 15.29 (4.027)
  AST, Day 5: number analyzed (Participants) | 14 | 13
  AST, Day 5 | 16.29 (4.581) | 17.54 (11.230)
  CPK, Day -1 | 141.50 (106.360) | 121.36 (95.447)
  CPK, Day 5: number analyzed (Participants) | 14 | 13
  CPK, Day 5 | 75.71 (34.003) | 62.38 (20.077)

25. Secondary Outcome: Absolute Values of Clinical Chemistry Parameters: Direct Bilirubin, Total Bilirubin and Creatinine
Description: Blood samples were collected for analyzing absolute values of direct bilirubin, total bilirubin and Creatinine.
Time Frame: On Day -1 (admission) and Day 5 (Discharge)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Micromoles per liter
  Direct Bilirubin, Day -1 | 2.86 (1.562) | 3.57 (1.158)
  Direct Bilirubin, Day 5: number analyzed (Participants) | 14 | 13
  Direct Bilirubin, Day 5 | 3.14 (0.949) | 2.46 (1.391)
  Total Bilirubin, Day -1 | 9.64 (3.954) | 11.43 (3.877)
  Total Bilirubin, Day 5: number analyzed (Participants) | 14 | 13
  Total Bilirubin, Day 5 | 9.57 (2.709) | 8.08 (2.397)
  Creatinine, Day -1 | 63.36 (11.311) | 69.57 (12.145)
  Creatinine, Day 5: number analyzed (Participants) | 14 | 13
  Creatinine, Day 5 | 71.29 (12.363) | 61.77 (9.427)

26. Secondary Outcome: Absolute Values of Clinical Chemistry Parameter: Total Protein
Description: Blood samples were collected for analyzing absolute values of Total protein.
Time Frame: On Day -1 (admission) and Day 5 (Discharge)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Grams per liter
  Day -1 | 75.21 (3.886) | 73.93 (3.149)
  Day 5: number analyzed (Participants) | 14 | 13
  Day 5 | 68.57 (3.106) | 68.00 (2.121)

27. Secondary Outcome: Absolute Values for Chemistry Parameters: Calcium, Sodium, Potassium, Blood Urea Nitrogen (BUN)
Description: Blood samples were collected for analyzing absolute values of Calcium, Sodium, Potassium, Blood Urea Nitrogen.
Time Frame: On Day -1 (admission) and Day 5 (Discharge)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Millimoles per liter
  Calcium, Day -1 | 2.535 (0.0769) | 2.549 (0.0934)
  Calcium, Day 5: number analyzed (Participants) | 14 | 13
  Calcium, Day 5 | 2.466 (0.0756) | 2.442 (0.0893)
  Sodium, Day -1 | 140.07 (0.829) | 139.43 (1.742)
  Sodium, Day 5: number analyzed (Participants) | 14 | 13
  Sodium, Day 5 | 140.21 (1.188) | 139.69 (1.032)
  BUN, Day -1 | 4.81 (0.903) | 4.96 (1.709)
  BUN, Day 5: number analyzed (Participants) | 14 | 13
  BUN, Day 5 | 4.66 (1.203) | 4.38 (0.791)

28. Secondary Outcome: Absolute Values for Chemistry Parameter: Glucose
Description: Blood samples were collected for analyzing absolute values of glucose.
Time Frame: Baseline (Pre-dose at Day 1 and Day 4); 0.25, 0.5, 1 hour (h), 1.5 h, 2 h, 4 h post-dose at Day 1 and Day 4
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Millimoles per liter
  Baseline (Day 1, Predose) | 5.04 (0.599) | 4.89 (0.297)
  Day 1, 15 min post-dose | 5.43 (2.067) | 5.02 (0.587)
  Day 1, 30 min post-dose | 5.64 (1.790) | 5.14 (0.482)
  Day 1, 1 h post-dose | 5.47 (1.221) | 5.24 (0.533)
  Day 1, 1.5 h post-dose | 5.44 (0.925) | 5.11 (0.369)
  Day 1, 2 h post-dose | 5.24 (0.626) | 4.90 (0.335)
  Day 1, 4 h post-dose | 4.74 (0.378) | 4.71 (0.348)
  Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  Baseline (Day 4, Predose) | 4.76 (0.290) | 5.03 (0.964)
  Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 15 min post-dose | 5.06 (0.838) | 5.24 (2.514)
  Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 30 min post-dose | 5.13 (0.637) | 5.34 (2.064)
  Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 1 h post-dose | 5.15 (0.455) | 5.33 (1.434)
  Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 1.5 h post-dose | 5.11 (0.296) | 5.24 (1.171)
  Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 2 h post-dose | 4.96 (0.262) | 5.11 (0.999)
  Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 4 h post-dose | 4.71 (0.248) | 4.66 (0.380)

29. Secondary Outcome: Number of Participants With Urinalysis Parameters by Dipstick Method
Description: Urine samples were collected to assess glucose, ketones, occult blood, protein, urobilinogen and bilirubin by dipstick method. The dipstick test gave results in a semi-quantitative manner indicating proportional concentrations in the urine sample. Results are presented as'(+)' indicating 'equivocal', '+' indicating 'trace amount', '++' indicating 'positive', and 'negative'.
Time Frame: On Day -1 (admission) and Day 5 (Discharge)
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Participants
  Urine Protein, Day -1: (+) | 0 | 0
  Urine Protein, Day -1: + | 0 | 1
  Urine Protein, Day -1: ++ | 0 | 0
  Urine Protein, Day -1: Negative | 14 | 13
  Urine Protein, Day 5: number analyzed (Participants) | 14 | 13
  Urine Protein, Day 5: (+) | 0 | 0
  Urine Protein, Day 5: + | 0 | 1
  Urine Protein, Day 5: ++ | 0 | 0
  Urine Protein, Day 5: Negative | 14 | 12
  Urine Glucose, Day -1: (+) | 0 | 0
  Urine Glucose, Day -1: + | 0 | 0
  Urine Glucose, Day -1: ++ | 0 | 0
  Urine Glucose, Day -1: Negative | 14 | 14
  Urine Glucose, Day 5: number analyzed (Participants) | 14 | 13
  Urine Glucose, Day 5: (+) | 0 | 0
  Urine Glucose, Day 5: + | 0 | 0
  Urine Glucose, Day 5: ++ | 0 | 0
  Urine Glucose, Day 5: Negative | 14 | 13
  Ketones, Day -1: (+) | 0 | 0
  Ketones, Day -1: + | 0 | 0
  Ketones, Day -1: ++ | 0 | 0
  Ketones, Day -1: Negative | 14 | 14
  Ketones, Day 5: number analyzed (Participants) | 14 | 13
  Ketones, Day 5: (+) | 1 | 1
  Ketones, Day 5: + | 0 | 0
  Ketones, Day 5: ++ | 0 | 0
  Ketones, Day 5: Negative | 13 | 12
  Urine Hemoglobin, Day -1: (+) | 2 | 0
  Urine Hemoglobin, Day -1: + | 0 | 3
  Urine Hemoglobin, Day -1: ++ | 0 | 1
  Urine Hemoglobin, Day -1: Negative | 12 | 10
  Urine Hemoglobin, Day 5: number analyzed (Participants) | 14 | 13
  Urine Hemoglobin, Day 5: (+) | 2 | 1
  Urine Hemoglobin, Day 5: + | 0 | 0
  Urine Hemoglobin, Day 5: ++ | 0 | 0
  Urine Hemoglobin, Day 5: Negative | 12 | 12

30. Secondary Outcome: Absolute Values of Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Blood pressure measurements were assessed with a completely automated device after the participant has been resting for at least 5 minutes in the supine position. Manual techniques were used only if an automated device was not available.
Time Frame: Baseline (Pre-dose at Day 1 and Day 4); 0.25, 0.5, 1 hour (h), 1.5 h, 2 h, 4 h post-dose at Day 1 and Day 4
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury [mmHg]
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Millimeters of mercury [mmHg]
  DBP, Baseline (Day 1, Predose) | 69.1 (6.27) | 69.4 (7.21)
  DBP, Day 1, 15 min post-dose | 68.2 (6.42) | 67.8 (7.82)
  DBP, Day 1, 30 min post-dose | 70.6 (9.30) | 69.1 (9.21)
  DBP, Day 1, 1 h post-dose | 67.8 (7.16) | 67.4 (8.78)
  DBP, Day 1, 1.5 h post-dose | 65.3 (5.98) | 67.8 (8.46)
  DBP, Day 1, 2 h post-dose | 66.3 (4.18) | 66.1 (8.23)
  DBP, Day 1, 4 h post-dose | 68.1 (6.44) | 67.6 (8.99)
  DBP, Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  DBP, Baseline (Day 4, Predose) | 72.1 (6.64) | 67.9 (5.51)
  DBP, Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  DBP, Day 4, 15 min post-dose | 67.4 (7.59) | 64.9 (4.33)
  DBP, Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  DBP, Day 4, 30 min post-dose | 67.0 (6.23) | 63.8 (4.44)
  DBP, Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  DBP, Day 4, 1 h post-dose | 68.5 (7.86) | 65.4 (3.69)
  DBP, Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  DBP, Day 4, 1.5 h post-dose | 67.4 (6.48) | 63.6 (5.17)
  DBP, Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  DBP, Day 4, 2 h post-dose | 67.9 (7.71) | 64.1 (5.78)
  DBP, Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  DBP, Day 4, 4 h post-dose | 68.5 (6.31) | 65.6 (6.13)
  SBP, Baseline (Day 1, Predose) | 111.9 (8.49) | 113.0 (10.24)
  SBP, Day 1, 15 min post-dose | 118.2 (9.00) | 119.1 (10.27)
  SBP, Day 1, 30 min post-dose | 121.6 (15.05) | 118.6 (10.48)
  SBP, Day 1, 1 h post-dose | 114.9 (9.14) | 116.7 (8.91)
  SBP, Day 1, 1.5 h post-dose | 110.1 (8.27) | 115.7 (10.36)
  SBP, Day 1, 2 h post-dose | 111.5 (8.54) | 112.9 (10.57)
  SBP, Day 1, 4 h post-dose | 112.5 (8.84) | 112.0 (10.91)
  SBP, Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  SBP, Baseline (Day 4, Predose) | 114.8 (8.31) | 108.6 (7.15)
  SBP, Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  SBP, Day 4, 15 min post-dose | 119.1 (9.68) | 116.1 (9.72)
  SBP, Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  SBP, Day 4, 30 min post-dose | 119.8 (10.96) | 112.5 (7.87)
  SBP, Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  SBP, Day 4, 1 h post-dose | 115.2 (8.74) | 111.6 (11.15)
  SBP, Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  SBP, Day 4, 1.5 h post-dose | 115.9 (12.07) | 109.2 (7.61)
  SBP, Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  SBP, Day 4, 2 h post-dose | 115.9 (11.84) | 108.2 (10.60)
  SBP, Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  SBP, Day 4, 4 h post-dose | 113.6 (11.04) | 108.9 (9.18)

31. Secondary Outcome: Absolute Values of Pulse Rate
Description: Pulse rate measurements were assessed with a completely automated device after the participant has been resting for at least 5 minutes in the supine position. Manual techniques were used only if an automated device was not available.
Time Frame: Baseline (Pre-dose at Day 1 and Day 4); 0.25, 0.5, 1 hour (h), 1.5 h, 2 h, 4 h post-dose at Day 1 and Day 4
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
Number analyzed (Participants) | 14 | 14
Beats per minute
  Baseline (Day 1, Predose) | 58.6 (9.43) | 61.7 (9.75)
  Day 1, 15 min post-dose | 70.8 (9.54) | 71.8 (11.43)
  Day 1, 30 min post-dose | 69.4 (9.04) | 73.5 (12.86)
  Day 1, 1 h post-dose | 65.9 (9.14) | 68.9 (12.89)
  Day 1, 1.5 h post-dose | 63.6 (8.32) | 67.1 (11.01)
  Day 1, 2 h post-dose | 60.1 (7.79) | 65.1 (11.46)
  Day 1, 4 h post-dose | 58.3 (8.07) | 64.6 (10.27)
  Baseline (Day 4, Predose): number analyzed (Participants) | 14 | 13
  Baseline (Day 4, Predose) | 60.8 (9.77) | 55.2 (8.23)
  Day 4, 15 min post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 15 min post-dose | 74.1 (10.81) | 69.9 (8.41)
  Day 4, 30 min post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 30 min post-dose | 71.2 (9.89) | 66.3 (8.26)
  Day 4, 1 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 1 h post-dose | 69.3 (10.09) | 64.2 (8.21)
  Day 4, 1.5 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 1.5 h post-dose | 66.1 (9.62) | 62.3 (7.66)
  Day 4, 2 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 2 h post-dose | 65.1 (9.29) | 60.5 (7.88)
  Day 4, 4 h post-dose: number analyzed (Participants) | 14 | 13
  Day 4, 4 h post-dose | 62.9 (9.11) | 58.2 (6.84)

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) were collected from signing of the ICF, and all Adverse Events (AEs) were collected from start of study treatment up to Day 5 (discharge).
Description: Safety population included all participants who received at least one dose of study treatment.
Arm/Group | Salbutamol HFA-152a MDI | Salbutamol HFA-134a MDI
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 6/28 | 8/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salbutamol HFA-152a MDI (N=28) | Salbutamol HFA-134a MDI (N=27)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 0 (0) | 2 (2)
Vessel puncture site bruise (General disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-02-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT05791565/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT05791565/SAP_001.pdf